CLINICAL TRIAL: NCT06479226
Title: Efficacy of Cetylpyridinium Chloride and Zinc Mouthwash in Reducing the Occurrence of Symptoms Associated With the Flu and Cold Season - a Randomized Clinical Trial
Brief Title: Effect of Mouthwash in Reducing the Symptoms Associated With Flu and Cold Viruses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRO-2022-04-FLU-REG-BZ-ZM
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Healthy
MeSH Terms: interventions — Cetylpyridinium; Zinc; Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Toothbrushing alone
- cetylpyridinium chloride (0.075%) and zinc alcohol free mouthwash (Experimental): Toothbrushing + mouthrinse
  Interventions: Drug: cetylpyridinium chloride (0.075%) and zinc alcohol free mouthwash

INTERVENTIONS:
Drug: cetylpyridinium chloride (0.075%) and zinc alcohol free mouthwash — mouthrinse
  Arms: cetylpyridinium chloride (0.075%) and zinc alcohol free mouthwash

SUMMARY:
The aim of this study will be to evaluate the efficacy of regular cleaning of the oropharynx (via gargling) on the incidence of symptoms associated with flu and colds. The working hypothesis is that there will be a significant reduction in symptoms associated with flu and colds after using the mouthwash product, compared to the experimental control regime. A total of 150 individuals will be randomized to one of the two experimental regimens and followed for a period of 90 days. The experimental regimen consists of toothbrushing followed by gargling with a cetylpyridinium chloride (CPC) (0.075%) and zinc containing alcohol free rinse and the control regimen consists of toothbrushing alone. Participants will be instructed to brush their teeth twice a day for two minutes. Those allocated to the test regime will gargle with 20 ml of the mouthwash after each brushing. At the initial visit, participants will receive the products and instructions for use, as well as a daily log questionnaire. Participants will be asked to send their daily records once a week, using a messaging application. The proportion of days without any of the evaluated symptoms will be used as the main outcome. In addition, soft and hard tissue exams will be performed at the initial consultation, after 30 and 90 days of follow-up by a blinded researcher. Potential adverse events will be collected throughout the study. The groups will be compared using the chi-square test and one-way analysis of variance (ANOVA) will be used to compare the treatment group symptom rates between groups. The significance level will be set at 95%.

ELIGIBILITY:
Inclusion Criteria:

* Good systemic general health as determined by study investigators; Availability of 90 days to participate in the study;

Exclusion Criteria:

1. Those participating in any other clinical study; 2. Pregnant or breastfeeding; 3. Presence a history of allergies to oral hygiene products, personal hygiene products, or their ingredients; 4. Have mouth irritation or use oral anesthetic sprays; 5. Have diabetes; 6. Be undergoing extensive dental treatment or oral surgery during the study; 7. Present immunocompromised (HIV, AIDS, immunosuppressive drug therapy); 8. Use complete dentures; 9. Do not have carpal tunnel syndrome or arthritis in the hands. 10. Participant who substantially fails to follow the required protocols; 11. Participant who fails to attend scheduled appointments; 12. Participant who is treated, during the study period, with medications that may interfere with the parameters being analyzed in the study; 13. Participant who is treated by a medical or dental service, and this may interfere with the parameters being analyzed in the study; 14. Participant who develops serious adverse reactions. 15. The participant who chooses to terminate their participation in the study; 16. Participant reports being pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Upper Respiratory Symptom | 90 days
  any upper respiratory system associated with colds and flu according to the Wisconsin Upper Respiratory Symptom Survey (WURSS-21) Daily Symptom Report.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Muniz FWMG, Casarin M, Pola NM, Rosing CK, Silveira TMD, Silva FH, de Holanda GA, de Oliveira LV, Dantas PPA, Stewart B, Malheiros Z, Benitez C, Schaeffer L. Efficacy of regular gargling with a cetylpyridinium chloride plus zinc containing mouthwash can reduce upper respiratory symptoms. PLoS One. 2025 Feb 26;20(2):e0316807. doi: 10.1371/journal.pone.0316807. eCollection 2025. PMID 40009628